CLINICAL TRIAL: NCT06000436
Title: The Effect on Risk Awareness, Perception and Risk Factors of Motivational Interview-Based Cardiovascular Risk Reduction Program (CARDIOREP) in Taxi-Minibus Drivers: A Randomized Controlled Research
Brief Title: Cardiovascular Disease Risk of Awareness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serdar ulak, lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NecmettinEU70
Record Dates: First submitted 2023-07-19; First posted 2023-08-21 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/treatment (Experimental): Health education, mobile applications, monitoring, Cardiovascular disease risk assessment
  Interventions: Other: Cardiovascular disease risk assessment; Other: Training and Consultancy; Other: Mobile Application; Other: Monitoring
- Active group (Active Comparator): Cardiovascular disease risk assessment
  Interventions: Other: Cardiovascular disease risk assessment; Other: Monitoring

INTERVENTIONS:
Other: Cardiovascular disease risk assessment — Cardiovascular disease risk assessment
  Training and Consultancy Based on the literature, the researcher prepared a Training Guide for the Prevention of Cardiovascular Diseases, including the subjects of Cardiovascular Diseases and Risk Factors, Physical Activity, Smoking and Heart Health, BMI and Heart Health, Nutrition, and Stress. By using the training guide, training time for individual training intervention will be planned for one day of the week with the participants. Individual training will last 30 minutes at the stops with waiting areas during the working hours of the participants.
  Mobile Application To the participants in the intervention group 2, 4. In the 6th and 6th weeks, text messages will be shared once a week to increase motivation and prevent cardiovascular diseases.
  Monitoring Daily data from the previous week (cardio score, number of steps) will be taken from the Google Fit application.
Other: Training and Consultancy — Based on the literature, the researcher prepared a Training Guide for the Prevention of Cardiovascular Diseases, including the subjects of Cardiovascular Diseases and Risk Factors, Physical Activity, Smoking and Heart Health, BMI and Heart Health, Nutrition, and Stress. Using the training guide, training time for individual training intervention will be planned for one day of the week with the participants. Individual training will last 30 minutes at the stops with waiting areas during the participants' working hours.
  Arms: Intervention/treatment
Other: Mobile Application — To the participants in the intervention group 2, 4. In the 6th and 6th weeks, text messages will be shared once a week to increase motivation and prevent cardiovascular diseases.
  Text Messages Week 2 "Tobacco use causes 6 million deaths in the world. The risk of death is reduced by 90% in those who stop using tobacco. Alcohol use causes damage to the heart muscle, arrhythmia, and stroke. For a healthy life, you should stay away from smoking and alcohol. ' Week 4 '' Inadequate physical activity increases the risk of death from all causes. Physical activity reduces the risk of hypertension, stroke, and depression. 30 minutes of moderate-intensity physical activity daily is recommended.
  Week 6 "Adequate consumption of vegetables and fruits reduces the risk of cardiovascular disease. Saturated and trans fats increase the risk of cardiovascular disease. It is recommended to consume <5 g less per day to prevent cardiovascular diseases.
  Arms: Intervention/treatment
Other: Monitoring — Daily data from the previous week (cardio score, number of steps) will be taken from the Google Fit application.

SUMMARY:
The Cardiovascular Risk Reduction Program (CARDIOREP) aims to raise risk awareness and reduce risk factors.

DETAILED DESCRIPTION:
While 1/3 of premature deaths in individuals under the age of 70 in the world occur due to Cardiovascular Diseases (WHO 2022), circulatory system diseases are at the forefront with 36.76% according to the health statistics of the Ministry of Health in our country. It is necessary to raise awareness and gain healthy lifestyle behaviors in the prevention of cardiovascular diseases. The Cardiovascular Risk Reduction Program (CARDIOREP) aims to raise risk awareness and reduce risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Not having been diagnosed with cardiovascular disease.
* Using a smartphone.
* Agree to use the Google Fit App.

Exclusion Criteria:

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Disease Risk Awareness Rating Scale Scores | at the end of 0th, 6th, and 12th weeks
  The scale form consists of 3 sub-dimensions and 21 items. The sub-dimensions consist of perceived heart attack and stroke risk, healthy eating intentions, perceived benefits and intentions to change. A maximum score of 64 and a minimum score of 0 can be obtained from the scale. A higher score on the scale and its sub-dimensions indicates an increased awareness of cardiovascular diseases.

SECONDARY OUTCOMES:
Cardiovascular risk perception | at the end of 0th, 6th, and 12th weeks
  Perceived cardiovascular disease risk in the next 10 years is questioned as low, moderate, high and very high.
International Physical Activity Questionnaire Scores | at the end of 0th, 6th, and 12th weeks
  The international physical activity questionnaire (Short Form) consists of 7 questions. The questionnaire asks about the number of days of vigorous, moderate, mild physical activity in the last 7 days and how much of the day, and how much time is spent sitting in individuals who do not engage in physical activity. It provides the calculation of the energy expended by the activities in meters. A high score on the scale form indicates being active in physical activity.
Beck Anxiety Scale Scores | at the end of 0th, 6th, and 12th weeks
  The scale form consists of 21 questions on a 4-point Likert scale (0=none, 3=seriously) about anxiety symptoms in the last one week.
Cardiovascular disease risk factors | at the end of 0th, 6th, and 12th weeks
  anthropometric measurements weight (Kilograms)
Cardiovascular disease risk factors | at the end of 0th, 6th, and 12th weeks
  anthropometric measurements height (meter)
Cardiovascular disease risk factors | at the end of 0th, 6th, and 12th weeks
  anthropometric measurements hip circumference (centimeters)
Cardiovascular disease risk factors | at the end of 0th, 6th, and 12th weeks
  anthropometric measurements waist circumference (centimeters)
Cardiovascular disease risk factors | at the end of 0th, 6th, and 12th weeks
  blood pressure (mmHg)

IPD SHARING:
Plan to Share IPD: No